CLINICAL TRIAL: NCT02572830
Title: Blocking Memory Reconsolidation by Eye Movement Desensitization and Reprocessing (EMDR)
Brief Title: Reconsolidation and EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Christoph Müller-Pfeiffer, PD. Dr., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: F-86401-09-01
Record Dates: First submitted 2015-10-04; First posted 2015-10-09 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: PTSD
Keywords: Reconsolidation; EMDR; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Bilateral Eye Movements (Experimental): Delayed Bilateral Eye Movements after reactivation of fear-memory.
  Interventions: Behavioral: Delayed Bilateral Eye Movements
- Undelayed Bilateral Eye Movements (Active Comparator): Undelayed Bilateral Eye Movements after reactivation of fear-memory.
  Interventions: Behavioral: Undelayed Bilateral Eye Movement

INTERVENTIONS:
Behavioral: Delayed Bilateral Eye Movements — Bilateral Eye Movements followed by a 10 min delay after reactivation of fear-memory.
  Arms: Delayed Bilateral Eye Movements
Behavioral: Undelayed Bilateral Eye Movement — Bilateral Eye Movements followed by no delay after reactivation of fear-memory. reactivation of the fear memory trace during which the reactivated memory is assumed to be in a labile state.
  Arms: Undelayed Bilateral Eye Movements

SUMMARY:
Blocking of reconsolidation by pharmacological or behavioral means offers the therapeutic possibility of weakening traumatic memories in posttraumatic stress disorder (PTSD). Two reconsolidation-based interventions, propranolol and extinction learning, have been shown to weaken fear memories in human healthy subjects. However, the success of these interventions seems to be limited to weak conditioned fear memories. This calls for new, potentially more efficacious, interventions to be tested. Bilateral eye movements seem to be a promising candidate intervention for blocking reconsolidation due to the compelling evidence of Eye Movement Desensitization and Reprocessing as effective treatment in PTSD. The investigators' aim is to test bilateral eye movements as an active reconsolidation-blocking intervention in an optimized differential fear conditioning procedure that the investigators have recently developed. This novel experimental assay creates stronger fear memories in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 years and 60 years of age
* Presence of a manageable, nonphobic fear of spiders as determined by scores above the mean (male: 8.06; female: 10.46) on the German adapted Spider Phobia Questionnaire (SPQ; 38) and phobia criteria extracted from the Structured Clinical Interview for DSM-5 Axis I Disorders (SCID-I; 39)
* Signed Informed Consent after being informed

Exclusion Criteria:

* Current or past neurological or other medical condition affecting the brain
* Current use of any medication (except contraceptives, herbal medicine)
* Known or suspected non-compliance, drug or alcohol misuse
* Presence of any current psychiatric disorders determined by the Mini International Neuropsychiatric Interview (MINI; 40)
* Inability to follow the procedures of the study, e.g. due to language problems
* No SC response to physical (Valsalva maneuver), psychological (mental arithmetic) and/or auditive (handclapping) stressor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-07 (Actual)

PRIMARY OUTCOMES:
Skin conductance (SC) response | Change from Day 1 (acquisition) fear conditioned SC response at day 3 (testing of renewal, reinstatement) and day 30 follow-up (testing of spontaneous recovery/renewal, savings)

SECONDARY OUTCOMES:
Blood oxygenation level dependent (BOLD) response | Change from Day 1 (acquisition) fear conditioned BOLD response at day 3 (testing of renewal, reinstatement) and day 30 follow-up (testing of spontaneous recovery/renewal, savings)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mueller-Pfeiffer, MD, Principal Investigator — University Hospital of Zurich, Department of Psychiatry and Psychotherapy
Locations (1):
- University Hospital Zurich, Department of Psychiatry and Psychotherapy, Zurich, Canton of Zurich, Switzerland